CLINICAL TRIAL: NCT01710319
Title: Mechanisms of Immunosurveillance for Lung Cancer
Acronym: MechLungCa
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Saint Louis VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 201110275
Record Dates: First submitted 2012-10-11; First posted 2012-10-19 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: Immunoregulation; Natural Killer Cells
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood draw will be obtained from patients in order to complete flow cytometry to analyze NK-specific markers to determine NK cell abundance and phenotypic expression. Obtain an optional blood draw on pts at least 30 days from the initial draw if transient confounders (viral infections or leukemoid reactions-a benign transient post-viral increase in WBCs) noted that could affect the NK Cell's behavior and interfere with the results.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- smoker with lung cancer: patients that smoke greater than 45 pack years or have end organ damage due to cigarette smoking and have lung cancer
  Interventions: Other: blood draw
- smoker without lung cancer: patients that smoke greater than 45 pack years or have end organ damage due to cigarette smoking and do not have lung cancer
  Interventions: Other: blood draw
- nonsmoker with lung cancer: patients that have smoked less than 100 cigarettes in their lifetime and have lung cancer
  Interventions: Other: blood draw
- nonsmoker without lung cancer: patients that have smoked less than 100 cigarettes in their lifetime and do not have lung cancer
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — a blood specimen will be obtained from each patient in the four groups. An optional blood draw after 30 days of initial blood specimen if indicated.

SUMMARY:
The purpose of this research study is to investigate the differences in "natural killer (NK) blood cells, a type of white blood cell that fights infection in the body, among different types of patients that have lung surgery. The four different groups of patients are:

* smokers with lung cancer
* smokers without lung cancer
* non-smokers with lung cancer
* non-smokers without lung cancer.

DETAILED DESCRIPTION:
Research has shown that different strains of mice possess varying susceptibility to lung cancer. C3H and C57BL6 mice are highly resistant to lung cancer, whereas A/J and 129 mice are very susceptible to lung cancer. Data from our lab shows that the mice have different numbers of natural killer (NK) cells as well as different characteristics of those cells. C3H and C57BL6 mice have higher numbers of NK cells as well as higher expression of CD11b, whereas A/J and 129 mice have lower numbers and lower expression.

These findings justify parallel investigation of NK cells in human populations resistant and susceptible to lung cancer. Through blood samples, circulating NK cells can be counted and phenotypically analyzed. Smoking can be used as a factor to establish lung cancer risk. Additionally, non-smokers suffering from lung cancer provide an opportunity to investigate whether lung cancer patients have lower abundance of NK cells and lesser expression of CD11b, independent of the effects of smoking.

Objective:

The main goal of this study is to investigate the quantitative and phenotypic differences in circulating NK cells among human populations. Participants will be classified as heavy smokers (HS), non-smokers (NS), those suffering from lung cancer (LC), and those free from lung cancer (NC).

Hypothesis #1: NS/LC participants will have fewer NK cells and lower expression of CD11b compared to HS/NC and NS/NC participants.

Hypothesis #2: NS/LC participants will have more numerous NK cells and higher expression of CD11b compared to HS/LC participants.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater to 18 years
* Ability to read and write in English
* Able to participate in the informed consent process

Exclusion Criteria:

* Known active hepatitis B, hepatitis C, or HIV/AIDs (found in medical record)
* Chemotherapy or radiation therapy within 3 months of enrollment
* Type 1 Diabetes Mellitus
* Rheumatoid arthritis, Lupus, Multiple Sclerosis, or any other autoimmune disease as deemed necessary for exclusion by the Principal Investigator
* Previous organ transplant
* Blood transfusion within 3 months prior to enrollment
* Any previous cancer, excluding a previous lung cancer
* Steroid use within 4 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be patients that visit the Thoracic Surgery clinic or healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2012-09; Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
Number of NK cells | Within 5 minutes of blood arrival to lab, processing begins and blood is frozen. Flow cytometry will be completed 1 to 3 months after blood is frozen. Data presentation in 1 to 2 years.
  The first outcome measure is the determination of the number of NK cells as a percentage of all CD45+cells.

SECONDARY OUTCOMES:
Expression of CD11b | Within 5 minutes of blood arrival to the lab, processing begins and blood is frozen. Flow cytometry will be completed 1 to 3 months after blood is frozen. Data presentation in 1 to 2 years.
  Expression of CD11b determined by flow cytometry as compared to control (nonsmoker/no cancer cohort. Flow cytometry will be used to analyze NK-specific markers in the blood samples to determine NK cell abundance and phenotypic expression. The NS/NC cohort will serve as the control for measuring CD11b expression.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Krupnick, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Bach PB, Kattan MW, Thornquist MD, Kris MG, Tate RC, Barnett MJ, Hsieh LJ, Begg CB. Variations in lung cancer risk among smokers. J Natl Cancer Inst. 2003 Mar 19;95(6):470-8. doi: 10.1093/jnci/95.6.470. PMID 12644540
- [Background] Bondy SJ, Victor JC, Diemert LM. Origin and use of the 100 cigarette criterion in tobacco surveys. Tob Control. 2009 Aug;18(4):317-23. doi: 10.1136/tc.2008.027276. Epub 2009 Jun 1. PMID 19491091
- [Background] Murala SS, Gelman AE, Kreisel D, Krupnick AS. Natural killer cells play a critical role in immunosurveillance for murine lung cancer. American Surgical Congress, Proceedings in The Journal of Surgical Research 2011; 165: 292-293.